CLINICAL TRIAL: NCT07102329
Title: THE REAL-LIFE BURDEN OF ESOPHAGEAL CANCER IN EOSINOPHILIC ESOPHAGITIS: A COMPARATIVE PROPENSITY-MATCHED ANALYSIS FROM A GLOBAL MULTICENTER DATABASE (THE ESCAPE STUDY)
Brief Title: BURDEN OF ESOPHAGEAL CANCER IN EOSINOPHILIC ESOPHAGITIS (ESCAPE STUDY)
Acronym: ESCAPE
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Collaborators: TriNetX, LLC (Unknown); Vita-Salute San Raffaele University (Unknown)
Responsible Party: Principal Investigator, Alberto Barchi, Medical Doctor, IRCCS San Raffaele
Other Study IDs: ESCAPE-1
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Eosinophilic Esophagitis (EoE)
Keywords: Eosinophilic Esophagitis; Esophageal Cancer; Gastroesophageal Reflux Disease; Barrett Esophagus; Risk
MeSH Terms: conditions — Eosinophilic Esophagitis; Esophageal Neoplasms; Gastroesophageal Reflux; Barrett Esophagus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- A) primary cohort of EoE patients: The primary cohort of the main analysis was built to include all eosinophilic esophagitis (EoE) patients, therefore implementing the ICD-10 code specific for the disease (K20.0). In order not to include other eosinophilic gastrointestinal disorders (EGIDs) primary cohort was built excluding the following ICD-10(ICD-9) codes:
  * K52.81: Eosinophilic Gastritis or Gastroenteritis
  * K52.82: Eosinophilic Colitis
  * K558.4: Eosinophilic gastroenteritis and colitis
  Following diagnosis were excluded if happened on or before the index event:
  * ICD-10-K22.7 Barrett Esophagus
  * ICD-10-K22.71 Barrett Esophagus with dysplasia
  * ICD-10-K22.711 Barrett Esophagus with high-grade dysplasia
  * ICD-10-K22.719 Barrett Esophagus with dysplasia, unspecified
  * ICD-10-K22.710 Barrett Esophagus with low-grade dysplasia
  * ICD-10-K22.1 Ulcer of the esophagus
  * ICD-10-K22.10 Ulcer of the esophagus without bleeding
  * ICD-10-K22.11 Ulcer of the esophagus with bleeding
  * ICD-10-C15 Esophageal cancer
- Cohort B: Pure EoE without BE/GERD: The secondary cohort (Cohort B) of the main analysis was built to include all eosinophilic esophagitis (EoE) patients, therefore implementing the ICD-10 code specific for the disease (K20.0). In order not to include other eosinophilic gastrointestinal disorders (EGIDs) leading to confounding clinical profiles, this primary cohort was built excluding the following ICD-10(ICD-9) codes:
  * K52.81: Eosinophilic Gastritis or Gastroenteritis
  * K52.82: Eosinophilic Colitis
  * K558.4: Eosinophilic gastroenteritis and colitis
  To eliminate the confounding effect of BE and objective GERD was built with the exclusion from cohort A of the following diagnosis:
  * ICD-10-K22.7 Barrett Esophagus
  * ICD-10-K22.71 Barrett Esophagus with dysplasia
  * ICD-10-K22.711 Barrett Esophagus with high-grade dysplasia
  * ICD-10-K22.719 Barrett Esophagus with dysplasia, unspecified
  * ICD-10-K22.710 Barrett Esophagus with low-grade dysplasia
  * ICD-10-K22.1 Ulcer of the esophagus
  * ICD-10-K22.11 Ulcer of the esophagus with bleeding
- Control group: The control group cohort was built in order to minimize the risk of selection bias, using the general code for "encounter for general examination without complaint, suspected or reported diagnosis" ICD-10 Z00 with the exclusion of the following codes related to EoE diagnosis (ICD10-K20.0). In order to minimize the overestimation of time-to-event risk of primary outcome, the following diagnosis were excluded if happened on or before the index event:
  * ICD-10-K22.7 Barrett Esophagus
  * ICD-10-K22.71 Barrett Esophagus with dysplasia
  * ICD-10-K22.711 Barrett Esophagus with high-grade dysplasia
  * ICD-10-K22.719 Barrett Esophagus with dysplasia, unspecified
  * ICD-10-K22.710 Barrett Esophagus with low-grade dysplasia
  * ICD-10-K22.1 Ulcer of the esophagus
  * ICD-10-K22.10 Ulcer of the esophagus without bleeding
  * ICD-10-K22.11 Ulcer of the esophagus with bleeding
  * ICD-10-C15 Esophageal cancer To restrict the number of patients in the control group only patients with an "ambulatory" encounter.

SUMMARY:
Eosinophilic esophagitis (EoE) is a chronic, immune-mediated inflammatory disorder of the esophagus that can lead to symptoms such as dysphagia and food impaction. In recent years, a potential association between EoE and esophageal cancer (EC) has been proposed, though evidence remains inconsistent and may be influenced by overlapping conditions like gastroesophageal reflux disease (GERD) and Barrett's esophagus (BE).

The purpose of this study was to determine whether patients with EoE are at increased risk of developing esophageal cancer, and to clarify whether any observed risk is intrinsic to EoE or instead related to coexisting GERD or BE.

The main research question was: Is eosinophilic esophagitis independently associated with an increased risk of esophageal cancer, or is this risk mediated by overlapping conditions such as GERD or Barrett's esophagus? To address this, we conducted a retrospective, multicenter cohort study using real-world data from TriNetX, a global federated health research network aggregating electronic medical records from approximately 100 million patients.

DETAILED DESCRIPTION:
Eosinophilic esophagitis (EoE) is a chronic, immune-mediated inflammatory disease of the esophagus, often presenting with symptoms such as dysphagia and food impaction. Recent literature has raised concerns about a potential association between EoE and the development of esophageal cancer (EC), though findings are inconsistent and possibly confounded by coexisting gastroesophageal reflux disease (GERD) or Barrett's esophagus (BE).

The objective of this study was to assess whether EoE independently increases the risk of esophageal cancer, or whether any observed risk is primarily driven by overlapping conditions such as GERD or BE.

This was a retrospective, multicenter cohort study utilizing TriNetX, a global federated health research network that provides access to real-world data from electronic medical records (EMRs) of over 100 million patients across more than 100 large healthcare organizations (HCOs), predominantly located in the United States. The network supports cohort design, real-time analytics, and privacy-preserving analytics within a federated data environment.

Patients were selected based on the ICD-10 diagnosis code for eosinophilic esophagitis (K20.0) recorded between January 1, 2000, and March 31, 2025. To isolate the specific contribution of EoE to cancer risk, two distinct EoE cohorts were defined:

Cohort A: All patients with a diagnosis of EoE, excluding only other eosinophilic gastrointestinal disorders (EGIDs), thereby including individuals with coexisting GERD or BE Cohort B: A more stringently defined "pure EoE" group, excluding patients with any diagnosis of GERD, BE, or other EGIDs, in order to assess the cancer risk attributable to EoE in isolation.

Each EoE cohort was compared to a control cohort comprising patients who had outpatient encounters for non-specific or undefined reasons (ICD-10 Z00), and who had no recorded diagnosis of EoE and any instance of EC or BE before the index event.

To reduce bias and account for confounding factors, a 1:1 propensity score matching was performed using a nearest-neighbor greedy algorithm, with several matching variables.

Time-to-event analysis was designed using Kaplan-Meier survival curves, with censoring applied at the last clinical encounter. Comparative analysis of cancer incidence between groups was planned through log-rank testing, and both hazard ratios (HRs) and risk differences (RDs) were to be calculated.

This study design aims to provide a clearer understanding of whether EoE itself constitutes an independent risk factor for esophageal cancer, after accounting for potential confounding conditions.

ELIGIBILITY:
Inclusion Criteria:

* EoE diagnosed patients according to ICD-10 code K20

Exclusion Criteria:

* Patients diagnosed with other EGIDs (- K52.81: Eosinophilic Gastritis or Gastroenteritis
* K52.82: Eosinophilic Colitis
* K558.4: Eosinophilic gastroenteritis and colitis)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: - EoE diagnosed patients according to ICD-10 code K20, compared to control population
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2025-07-23 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Hazard Ratio (HR) of esophageal cancer (EC) in EoE cohort A versus controls | from January 2000 to July 2025
  Hazard ratios (HRs) and 95% confidence intervals (CIs) for EC development in cohort A versus controls, derived from Cox proportional hazards models, where cohort assignment served as the primary covariate. The proportional hazards assumption was evaluated using the generalized Schoenfeld residuals method.

SECONDARY OUTCOMES:
Hazard Ratio (HR) of esophageal cancer (EC) in EoE cohort B versus controls | From January 2000 to July 2025
  Hazard ratios (HRs) and 95% confidence intervals (CIs) for EC development in cohort A versus controls, derived from Cox proportional hazards models, where cohort assignment served as the primary covariate. The proportional hazards assumption was evaluated using the generalized Schoenfeld residuals method.
  Secondary analysis in order to extract the real estimate of having EC in pure EoE versus controls.
Hazard Ratio (HR) of adenocarcinoma (EAC) or squamous cell carcijoma (SCC in EoE cohort A versus controls | from January 2000 to July 2025
  Hazard ratios (HRs) and 95% confidence intervals (CIs) for EAC vs SCC development in cohort A versus controls, derived from Cox proportional hazards models, where cohort assignment served as the primary covariate. The proportional hazards assumption was evaluated using the generalized Schoenfeld residuals method.
Hazard Ratio (HR) of adenocarcinoma (EAC) or squamous cell carcijoma (SCC in pure EoE cohort B versus controls | from January 2000 to July 2025
  Hazard ratios (HRs) and 95% confidence intervals (CIs) for EAC vs SCC development in cohort B versus controls, derived from Cox proportional hazards models, where cohort assignment served as the primary covariate. The proportional hazards assumption was evaluated using the generalized Schoenfeld residuals method.

OTHER OUTCOMES:
Hazard Ratio (HR) and Risk Difference (RD) of EC, SCC and EAC in cohort A vs cohort B | from January 2000 to July 2025
  Hazard ratios (HRs), risk difference (RD) and 95% confidence intervals (CIs) for EC vs EAC vs SCC development in cohort A versus cohort B (to further explore the impact of GERD/BE), derived from Cox proportional hazards models, where cohort assignment served as the primary covariate. The proportional hazards assumption was evaluated using the generalized Schoenfeld residuals method.
Estimate the incidence, prevalence proportion (/100,000 persons) and incidence rate (100,000 persons/year) for EC overall, EAC and SCC in cohort A and cohort B | from January 2000 to July 2025
  Estimate the incidence, prevalence proportion (/100,000 persons) and incidence rate (100,000 persons/year) for EC overall, EAC and SCC in cohort A and cohort B to highlight epidemiology data of cancer in the two EOE cohort to further delineate differences.
Estimate the incidence, prevalence proportion (/100,000 persons) and incidence rate (100,000 persons/year) for GERD and BE in cohort A | from January 2000 to July 2025
  Estimate the incidence, prevalence proportion (/100,000 persons) and incidence rate (100,000 persons/year) for GERD and BE in cohort A to appreciate the overall burden of GERD and BE in patients diagnosed with EoE

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Barchi, MD, Principal Investigator — IRCCS San Raffaele Hospital
Locations (1):
- IRCCS San Raffaele Hospital, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
No IPD used